CLINICAL TRIAL: NCT01105897
Title: Incidence of Deeply Infiltrating Endometriosis in Surgically Treated Endometriosis Patients and Long-term Results of Surgical Treatment in Terms of Pain, Quality of Life and Sexual Functioning
Brief Title: Prospective Study of the Outcomes of the Surgical Treatment of Deeply Infiltrating Endometriosis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: PaijatHame Central Hospital (Other)
Responsible Party: Principal Investigator, Marjaleena Setala, M.D., PaijatHame Central Hospital
Other Study IDs: ETLQ62/81
Record Dates: First submitted 2010-04-15; First posted 2010-04-19 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Endometriosis
Keywords: endometriosis; deep endometriosis; surgery; laparoscopy; chronic pain; quality of life; sexual function; complications; recurrence
MeSH Terms: conditions — Endometriosis; Chronic Pain; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgically treated endometriosis patients: Women scheduled for operation on suspected endometriosis in two study hospitals specialized in the surgical treatment of endometriosis between January 2005 - December 2007 (Päijät-Häme Central Hospital) and January 2008 - December 2008 (Helsinki University Hospital).
  Interventions: Procedure: Endometriosis surgery

INTERVENTIONS:
Procedure: Endometriosis surgery — Complete surgical excision of all visible endometriosis by multidisciplinary approach

SUMMARY:
The aim of this study is to examine the incidence of deeply infiltrating endometriotic lesions among surgically treated endometriosis patients, and examine the impact of endometriosis, and its surgical treatment, on severity of pain symptoms, quality of life, and sexual functioning.

DETAILED DESCRIPTION:
Patients scheduled for operation on suspected endometriosis in two study hospitals specialized in the surgical treatment of endometriosis between January 2005 - December 2007 (Päijät-Häme Central Hospital) and January 2008 - December 2008 (Helsinki University Hospital) were enrolled to the study. The diagnosis of endometriosis was histologically verified for all patients. Background data was collected from patients' age, body mass index, previous deliveries, previous endometriosis surgery, and current hormonal treatment for endometriosis.

From the beginning of January 2006 patients also completed preoperative questionnaires considering visual analogue scales (VAS) for pain symptoms (dysmenorrhea, deep dyspareunia, pain with urination and defecation, chronic pelvic pain, pain with ovulation), functional bowel and urinary symptoms, and 15D Quality of Life questionnaire, McCoy sexual functioning questionnaire, EHP-5 Short Form Endometriosis Profile questionnaire. Same questionnaires will also be completed six months, one year, two years, four years, and six years after the endometriosis operation. Follow-up questionnaires also contain questions concerning complications related to surgery, endometriosis recurrence, pregnancies, and infertility treatments.

ELIGIBILITY:
Inclusion Criteria:

* Finnish speaking patients scheduled for operation on suspected endometriosis

Exclusion Criteria:

* Non-Finnish speaking patients
* Previous hysterectomy.
* Previous bilateral salpingo-oophorectomy
* Any cancer
* Chronic inflammatory bowel or bladder disease
* Diabetes treated with insulin
* Rheumatoid arthritis.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women scheduled for operation on suspected endometriosis in two study hospitals between January 2005 - December 2007 (Päijät-Häme Central Hospital) and January 2008 - December 2008 (Helsinki University Hospital).
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2005-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Endometriosis related pain symptoms before, and one year after the endometriosis surgery | 12 months
  Endometriosis related pain symptoms (dysmenorrhea, deep dyspareunia, pain with urination and defecation, chronic pelvic pain, pain with ovulation) assessed with visual analogue scales (VAS) and measured before, six months and one year after the surgery.
The incidence of deeply infiltrating lesions among surgically treated endometriosis patients. | 3 years
  The incidence of deeply infiltrating endometriosis among consecutive patients operated on suspected endometriosis between January 2005- December 2007
Quality of life before, and one year after the endometriosis surgery | one year
  Quality of life assessed with 15D Quality of Life questionnaire and EHP-5 Short Form Endometriosis Profile questionnaire before the operation and, one year after the surgery.
Sexual functioning of endometriosis patients before, and one year after the surgery | one year
  Sexual functioning measured with McCoy sexual functioning questionnaire before and one year after the surgery.
Complication related to surgical treatment of deeply infiltrating endometriosis with one year postoperative follow-up | one year
  Prospective monitoring of intraoperative complications, complications during the hospital stay, and mailed questionnaires six months, and one year after the endometriosis operation containing questions concerning complications related to surgery.

SECONDARY OUTCOMES:
Recurrence of endometriosis after surgical treatment | six years
  Mailed questionnaires six months, one year, two years, four years, and six years after the surgical treatment of endometriosis containing questions about the recurrence of pain symptoms and about further endometriosis operations

CONTACTS AND LOCATIONS:
Overall Officials: Marjaleena Setälä, MD, Principal Investigator — Päijänne Tavastia Central Hospital; Jyrki Kössi, MD, PhD, Study Director — Päijänne Tavastia Central Hospital; Juha Mäkinen, Prof., Study Director — Turku University Hospital, Turku, Finland
Locations (1):
- Päijät-Häme Central Hospital, Lahti, Lahti, Finland

REFERENCES:
- [Background] Setälä M, Härkki P, Suvitie P, Fraser J, Jalkanen J, Kössi J, Perheentupa A, Mäkinen J. Is the presence of endometrioma always associated with more severe disease? Gynecol Surg, 2011 Jan. Epub ahead of print.
- [Background] Huhtinen K, Suvitie P, Hiissa J, Junnila J, Huvila J, Kujari H, Setala M, Harkki P, Jalkanen J, Fraser J, Makinen J, Auranen A, Poutanen M, Perheentupa A. Serum HE4 concentration differentiates malignant ovarian tumours from ovarian endometriotic cysts. Br J Cancer. 2009 Apr 21;100(8):1315-9. doi: 10.1038/sj.bjc.6605011. Epub 2009 Mar 31. PMID 19337252
- [Result] Kossi J, Setala M, Enholm B, Luostarinen M. The early outcome of laparoscopic sigmoid and rectal resection for endometriosis. Colorectal Dis. 2010 Mar;12(3):232-5. doi: 10.1111/j.1463-1318.2009.01923.x. Epub 2009 Apr 27. PMID 19438891
- [Result] Setala M, Savolainen H, Kossi J, Ranta T, Makinen J. Deeply infiltrating disease in surgically treated endometriosis patients. Acta Obstet Gynecol Scand. 2011 May;90(5):468-72. doi: 10.1111/j.1600-0412.2011.01097.x. Epub 2011 Mar 29. PMID 21314818
- [Result] Setala M, Kossi J, Silventoinen S, Makinen J. The impact of deep disease on surgical treatment of endometriosis. Eur J Obstet Gynecol Reprod Biol. 2011 Oct;158(2):289-93. doi: 10.1016/j.ejogrb.2011.04.046. Epub 2011 May 31. PMID 21621895
- [Result] Kossi J, Setala M, Makinen J, Harkki P, Luostarinen M. Quality of life and sexual function 1 year after laparoscopic rectosigmoid resection for endometriosis. Colorectal Dis. 2013 Jan;15(1):102-8. doi: 10.1111/j.1463-1318.2012.03111.x. PMID 22642851
- [Result] Setala M, Harkki P, Matomaki J, Makinen J, Kossi J. Sexual functioning, quality of life and pelvic pain 12 months after endometriosis surgery including vaginal resection. Acta Obstet Gynecol Scand. 2012 Jun;91(6):692-8. doi: 10.1111/j.1600-0412.2012.01394.x. Epub 2012 Apr 30. PMID 22404128